CLINICAL TRIAL: NCT03381521
Title: The Clinical Volume Effect of Nerve Hydrodissection in Patients With Carpal Tunnel Syndrome
Brief Title: The Volume Effect of Nerve Hydrodissection for Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Yung-Tsan Wu, Attending Physician of Department of Physical Medicine and Rehabilitation, Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Nerve hydrodissection for CTS
Record Dates: First submitted 2017-12-18; First posted 2017-12-22 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Carpal Tunnel Syndrome
Keywords: nerve hydrodissection
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Ultrasonography; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Ultrasound-guided nerve hydrodissection with 10cc normal saline
  Interventions: Procedure: Ultrasound-guided nerve hydrodissection; Device: Ultrasound; Drug: Normal saline
- Group B (Active Comparator): Ultrasound-guided nerve hydrodissection with 5cc normal saline
  Interventions: Procedure: Ultrasound-guided nerve hydrodissection; Device: Ultrasound; Drug: Normal saline

INTERVENTIONS:
Procedure: Ultrasound-guided nerve hydrodissection — Ultrasound-guided nerve hydrodissection with 10cc normal saline between carpal tunnel and median nerve.
  Arms: Group A
Procedure: Ultrasound-guided nerve hydrodissection — Ultrasound-guided nerve hydrodissection with 5cc normal saline between carpal tunnel and median nerve.
  Arms: Group B
Device: Ultrasound — The ultrasound was used to measure cross-sectional area and injection guidance
Drug: Normal saline — The normal saline was used for injection solution

SUMMARY:
Carpal tunnel syndrome (CTS) is the most common peripheral entrapment neuropathy with involving compression of the median nerve in the carpal tunnel. Although many conservative managements of CTS, the effectiveness of these methods is insignificant or only persist for a short duration. The technique of nerve hydrodissection is now commonly used for peeling the nerve from surrounding soft tissue, which may help allow the impulse to pass, and rescue the nerve with ischemic damage. However, the exact effect and interval of hydrodissection are unknown because of the lack of well-designed studies Hence, investigators design a randomized, double- blind, controlled trail to assess the therapeutic effect of ultrasound-guided nerve hydrodissection in patients with CTS.

DETAILED DESCRIPTION:
After obtaining written informed consent, patients clinically diagnosed with mild-to-moderate CTS were inclused and randomized into three groups. Group A, patients received one-session of ultrasoung-guided nerve hydrodissection with 10cc normal saline; Group B, patients received one-session of ultrasoung-guided nerve hydrodissection with 5cc normal saline; The injection syringe was covered to obscure the nature of its contents and patients were asked to turn their head away so that they would not see the procedure. As a result, patients were blinded to the treatment condition. The primary outcome is Boston Carpal Tunnel Syndrome Questionnaire (BCTQ) and secondary outcomes include visual analog scale (VAS), cross-sectional area (CSA) of the median nerve, sensory nerve conduction velocity of the median nerve, and global assessment of treatment. The evaluations were performed pretreatment as well as on the 2nd week, 1st, 3rd and 6th month after injecton.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20-80 year-old.
* Diagnosis was confirmed using an electrophysiological study

Exclusion Criteria:

* Cancer
* Coagulopathy
* Pregnancy
* Inflammation status
* Cervical radiculopathy
* Polyneuropathy, brachial plexopathy
* Thoracic outlet syndrome
* Previously undergone wrist surgery or steroid injection for CTS

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline of severity of symptoms and functional status on 2nd week, 1st, 3rd and 6th month after injection | Pre-treatment, 2nd week, 1st, 3rd and 6th month after injection
  Using the Boston Carpal Tunnel Syndrome Questionnaire (BCTQ) to measure the severity of symptoms and functional status before treatment and multiple time frame after treatment. BCTQ includes two subscale (11 questions in symptom severity and 8 questions in functional status). The scores ranged from 0 to 5 points in each question, in which zero score refered to as mildest and no difficulty in activity; five scores mean most worst severity and dysfunction.

SECONDARY OUTCOMES:
Change from baseline of pain on 2nd week, 1st, 3rd and 6th month after injection | Pre-treatment, 2nd week, 1st, 3rd and 6th month after injection
  Using the Visual analog scale (VAS) to measure the pain scale before treatment and multiple time frame after treatment. The VAS score range from 10 (tremendously harsh pain) to 0 points (no pain)
Change from baseline of cross-sectional area of the median nerve on 2nd week, 1st, 3rd and 6th month after injection | Pre-treatment, 2nd week, 1st, 3rd and 6th month after injection
  Using the musculoskeletal sonogram to measure the cross-sectional area of the median nerve before treatment and multiple time frame after treatment.
Change from baseline of conduction velocity, amplitude of median nerve on 2nd week, 1st, 3rd and 6th month after injection | Pre-treatment, 2nd week, 1st, 3rd and 6th month after injection
  Antidromic sensory nerve conduction velocity of the median nerve before treatment and multiple time frame after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Yung-Tsan Wu, MD, Principal Investigator — Department of Physical Medicine and Rehabilitation, Tri-Service General Hospital
Locations (1):
- Department of Physical Medicine and Rehabilitation, Tri-Service General Hospital, Taipei, Neihu District, Taiwan

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Wu YT, Ho TY, Chou YC, Ke MJ, Li TY, Tsai CK, Chen LC. Six-month Efficacy of Perineural Dextrose for Carpal Tunnel Syndrome: A Prospective, Randomized, Double-Blind, Controlled Trial. Mayo Clin Proc. 2017 Aug;92(8):1179-1189. doi: 10.1016/j.mayocp.2017.05.025. PMID 28778254
- [Result] Choi CK, Lee HS, Kwon JY, Lee WJ. Clinical implications of real-time visualized ultrasound-guided injection for the treatment of ulnar neuropathy at the elbow: a pilot study. Ann Rehabil Med. 2015 Apr;39(2):176-82. doi: 10.5535/arm.2015.39.2.176. Epub 2015 Apr 24. PMID 25932413
- [Result] Evers S, Thoreson AR, Smith J, Zhao C, Geske JR, Amadio PC. Ultrasound-guided hydrodissection decreases gliding resistance of the median nerve within the carpal tunnel. Muscle Nerve. 2018 Jan;57(1):25-32. doi: 10.1002/mus.25723. Epub 2017 Jul 6. PMID 28622409